CLINICAL TRIAL: NCT03466502
Title: Efficacy of Prophylactic Oral Vancomycin in Preventing Recurrent Clostridium Difficile Infection in Hospitalized Patients Requiring Antibiotics
Brief Title: Oral Vancomycin to Prevent Recurrent C Difficile Infection With Antibiotics
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Nevada, Reno (Other)
Collaborators: Renown Regional Medical Center (Other)
Responsible Party: Principal Investigator, Lauren Zion, PharmD, Pharmacist, University of Nevada, Reno
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1129396
Record Dates: First submitted 2018-03-08; First posted 2018-03-15 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Clostridium Difficile Infection
Keywords: vancomycin; Clostridium difficile; Clostridium difficile infection; Recurrent Clostridium difficile infection
MeSH Terms: conditions — Clostridium Infections | interventions — Vancomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- No oral vancomycin (No Intervention)
- Oral vancomycin 125 mg twice daily (Experimental)
  Interventions: Drug: Oral Vancomycin
- Oral vancomycin 125 mg daily (Experimental)
  Interventions: Drug: Oral Vancomycin

INTERVENTIONS:
Drug: Oral Vancomycin — Oral vancomycin will be given concurrently with antibiotics to hospitalized patients with a history of Clostridium difficile infection to prevent recurrence
  Arms: Oral vancomycin 125 mg daily; Oral vancomycin 125 mg twice daily

SUMMARY:
This study will assess the efficacy of oral vancomycin prophylaxis in preventing recurrent Clostridium difficile infection in hospitalized patients requiring oral or intravenous antibiotics for a suspected or confirmed bacterial infection.

DETAILED DESCRIPTION:
This study will assess the efficacy of oral vancomycin prophylaxis in preventing recurrent Clostridium difficile infection in hospitalized patients requiring oral or intravenous antibiotics for a suspected or confirmed bacterial infection.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Previous CDI diagnosis
3. Current admission with a suspected or a confirmed bacterial infection requiring antibiotics

Exclusion Criteria:

1. Active chronic diarrheal illness (eg, Crohn's disease, ulcerative colitis, short bowel syndrome)
2. Previous adverse reactions to oral vancomycin
3. Requiring metronidazole during hospitalization
4. Known pregnancy
5. Expected survival <72 hours
6. Patients receiving antibiotics only for surgical prophylaxis
7. Patients who received prophylactic oral vancomycin for the current antibiotic course prior to enrollment in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2018-03-08 (Actual); Primary Completion 2022-02-17 (Actual); Study Completion 2022-02-17 (Actual)

PRIMARY OUTCOMES:
Recurrent Clostridium difficile infection | During hospitalization or the 12 weeks after therapy
  Diarrheal illness, with at least 3 episodes of watery diarrhea over a 24 hour period and a positive toxin analysis or a positive PCR for Cdiff

SECONDARY OUTCOMES:
Recurrence rate of CDI according to C diff inducing properties of the prescribed antibiotics | During hospitalization or the 12 weeks after therapy
  * Low inducers: aminoglycosides, fosfomycin, glycopeptides, daptomycin, nitrofurantoin, linezolid, polymyxins, rifamycins, antifolates and/or sulfonamides, tetracyclines, tigecycline
  * Moderate inducers: penicillins, 1st generation cephalosporins, macrolides, azithromycin, streptogramins
  * High inducers: carbapenems, 2nd and greater generation cephalosporins, fluoroquinolones, clindamycin
Time between recurrent CDI and the last C diff infection | During hospitalization or the 12 weeks after therapy
Rate of recurrence of CDI in immunocompromised patients | During hospitalization or the 12 weeks after therapy
  HIV, Organ Transplantation, Current Immunosuppressive therapy, Hypogammaglobulinemia or steroids dose more than prednisone 20mg/day for 3 weeks
Rate of recurrence of CDI in patients with a history of the NAP-1 strain | During hospitalization or the 12 weeks after therapy
Rate of reported adverse events | During hospitalization or the 12 weeks after therapy
Mortality rate | During hospitalization or the 12 weeks after therapy

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Zion, PharmD, Principal Investigator — Renown Regional Medical Center
Locations (1):
- Renown Regional Medical Center, Reno, Nevada, United States

IPD SHARING:
Plan to Share IPD: No